CLINICAL TRIAL: NCT07322796
Title: Smoking Cessation Before Intervention in Patients With Pulmonary Nodules Requiring Further Diagnosis
Brief Title: Smoking Cessation Before Bronchoscopy or CT-guided Puncture
Status: Recruiting | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Jens Spießhöfer, PD Dr.Dr.med, RWTH Aachen University
Other Study IDs: 25-251
Record Dates: First submitted 2025-07-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Nodule, Solitary; Smoking Behaviors
Keywords: smoking; smoking cessation; pulmonary nodules
MeSH Terms: conditions — Solitary Pulmonary Nodule; Smoking; Smoking Cessation; Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smoking cessated: Patients who have stopped smoking since they were informed that they have a pulmonary lesion that needs clarification or after the diagnosis of cancer was communicated.
- Smoking not cessated: Patients who have not stopped smoking since they were informed that they have a pulmonary lesion that needs clarification or after the diagnosis of cancer was communicated.

SUMMARY:
Nicotine is the most common preventable cause of death and is responsible for over seven million deaths worldwide. If current trends continue, tobacco will kill more than eight million people worldwide every year by 2030. Smoking tobacco products is the most important risk factor for the development of lung cancer. Passive smoking is also a major cause of lung cancer. Since July 2024, smokers and former smokers have been able to receive a low-radiation CT scan under certain conditions to detect lung cancer at an early stage. It is therefore to be expected that the number of diagnoses of pulmonary lesions or nodules will increase in the near future. The risk of developing and dying from tobacco-related diseases is reduced once nicotine cessation begins. Screening all patients for tobacco use, e-cigarette use, and providing behavioral counseling and pharmacotherapy to quit smoking are among the most valuable preventive services we can offer in healthcare.

Nicotine dependence can be estimated using the so-called Fagerström test. An additional evaluation of nicotine behavior can be carried out by testing cotinine in urine, a method that is used, for example, in the listing for lung transplantation. Cotinine is a degradation product of nicotine that can be detected in the urine of smokers and passive smokers. Cotinine levels in urine depend on the frequency and quantity of nicotine consumption. The half-life of cotinine is 16 to 22 hours, which means that half of the cotinine is excreted from the body after this time. Another marker that can be used as a measure of tobacco consumption is carboxyhaemoglobin (COHb). This is hemoglobin with carbon monoxide at the binding site for oxygen. The reference range for carboxyhaemoglobin is 0.4 - 1.6 %. In smokers, values of 3-10 % are still considered normal.

In our department, the smoking status of patients is assessed upon first contact. Support options for smoking cessation are offered and, upon request, initiated. Previous studies have shown that smoking is a risk factor for complications after thoracic surgical procedures and that patients who underwent thoracic surgery quit smoking almost twice as often compared to patients who did not undergo surgery. However, to the best of our knowledge, there is currently no study regarding smoking cessation before intervention in patients with nodules needing clarification (bronchoscopy or CT-guided puncture).

Therefore, the aim of the study is to support and monitor smoking cessation before intervention in patients with nodules needing further diagnosis (bronchoscopy or CT-guided puncture).

DETAILED DESCRIPTION:
Patients who present to our outpatient clinic for the evaluation of a concerning round lesion (V1) are asked during the medical history taking whether they currently smoke. If the question is answered affirmatively, patients are urgently advised to quit smoking immediately. Support options for smoking cessation are presented, and if desired, a connection to a smoking cessation counseling program of the Federal Institute for Public Health ('rauchfrei ticket') is established. Furthermore, nicotine dependence is assessed using the Fagerström test, while COHb is determined through blood gas analysis and cotinine is measured in urine. During the planned result discussion (V2) after the inpatient stay for histological confirmation (either via bronchoscopy or CT-guided puncture), patients are asked if they have quit smoking and COHb and cotinine are measured again. After 3 months (V3), these values will be measured conclusively. In addition, the following data will be collected and documented from the patients: age, gender, height, weight, current medication, other illnesses, and current body plethysmography. Participation in the study does not change the course of the patients' stay in our clinic.

ELIGIBILITY:
Inclusion Criteria:

* The patient is an active smoker by the time of the initial presentation in our pneumological outpatient clinic for the clarification of a suspicious nodule

Exclusion Criteria:

* Current or past medically relevant illness or treatment that could affect the evaluability of the study.
* Expected lack of willingness to actively participate in study-related measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active smokers by the time of the initial presentation in our pneumological outpatient clinic for the clarification of a suspicious nodule
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Smoking Cessation | From enrollment to the end of the observation period 3 months later
  Patients who visit our outpatient clinic for the purpose of investigating a pulmonary lesion that requires clarification, are asked during the medical history if they are active smokers. If the answer is yes, patients are strongly advised to stop smoking immediately. Support options for smoking cessation are presented and, if desired, a connection to a smoking cessation counseling program offered by the Federal Institute for Public Health ("rauchfrei ticket") is established. In addition, nicotine dependence is assessed using the Fagerström test, COHb is determined by blood gas analysis, and cotinine is determined in urine. The same parameters will bei measured after 2-4 weeks and 3 months.
  As primary outcome measure, the number of patients who are likely to be smoke-free at the end of the observation period will be assessed.

SECONDARY OUTCOMES:
Analysis of demographic data | Within 3 months
  Age, gender, height, weight, comorbidities, medication
Spirometry (Lungfunction) | Within 3 Months
  During the study period, the spirometry of the enrolled patients will be assessed. The parameters that are included are the following:
  * peak expiratory flow (PEF) in L/s
  * mean expiratory flow at 75% of vital capacity (MEF75) in L/s
  * mean expiratory flow at 50% of vital capacity (MEF50) in L/s
  * mean expiratory flow at 25% of vital capacity (MEF25) in L/s
  * forced expiratory volume in 1 second (FEV1) in L
Bodyplethysmography (Lungfunction) | Within 3 months
  During the study period, the bodyplethysmography of the enrolled patients will be assessed. The parameters that are included are the following
  * total lung capacity (TLC) in L
  * vital capacity (VC) in L
  * residual volume (RV) in L
  * functional residual capacity assessed using plethysmography FRCpleth) in L
  * DLCO/VA [mmol/(min*kPa*L]
Diffusing capacity (lungfunction) | Within 3 months
  During the study period, the diffusing capacity of the enrolled patients will be assessed. The parameters that are included are the following
  - diffusing capacity of the lungs for carbon monoxide/aveolarventilation (DLCO/VA) in [mmol/(min*kPa*L]

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher Univ.-Prof. Dr.med, Study Director — University Hospital, Aachen
Locations (1):
- University RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mustoe MM, Clark JM, Huynh TT, Tong EK, Wolf TP, Brown LM, Cooke DT. Engagement and Effectiveness of a Smoking Cessation Quitline Intervention in a Thoracic Surgery Clinic. JAMA Surg. 2020 Sep 1;155(9):816-822. doi: 10.1001/jamasurg.2020.1915. PMID 32609348
- [Background] Wong C, Mohamad Asfia SKB, Myles PS, Cunningham J, Greenhalgh EM, Dean E, Doncovio S, Briggs L, Graves N, McCaffrey N. Smoking and Complications After Cancer Surgery: A Systematic Review and Meta-Analysis. JAMA Netw Open. 2025 Mar 3;8(3):e250295. doi: 10.1001/jamanetworkopen.2025.0295. PMID 40053349
- [Background] Marrufo AS, Kozower BD, Tancredi DJ, Nuno M, Cooke DT, Pollock BH, Romano PS, Brown LM. Thoracic Surgeons' Beliefs and Practices on Smoking Cessation Before Lung Resection. Ann Thorac Surg. 2019 May;107(5):1494-1499. doi: 10.1016/j.athoracsur.2018.11.055. Epub 2018 Dec 23. PMID 30586576
- [Background] Patnode CD, Henderson JT, Coppola EL, Melnikow J, Durbin S, Thomas RG. Interventions for Tobacco Cessation in Adults, Including Pregnant Persons: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2021 Jan 19;325(3):280-298. doi: 10.1001/jama.2020.23541. PMID 33464342
- [Background] Maciosek MV, Coffield AB, Edwards NM, Flottemesch TJ, Goodman MJ, Solberg LI. Priorities among effective clinical preventive services: results of a systematic review and analysis. Am J Prev Med. 2006 Jul;31(1):52-61. doi: 10.1016/j.amepre.2006.03.012. PMID 16777543
- [Background] Jha P, Ramasundarahettige C, Landsman V, Rostron B, Thun M, Anderson RN, McAfee T, Peto R. 21st-century hazards of smoking and benefits of cessation in the United States. N Engl J Med. 2013 Jan 24;368(4):341-50. doi: 10.1056/NEJMsa1211128. PMID 23343063
- [Background] Anthonisen NR, Skeans MA, Wise RA, Manfreda J, Kanner RE, Connett JE; Lung Health Study Research Group. The effects of a smoking cessation intervention on 14.5-year mortality: a randomized clinical trial. Ann Intern Med. 2005 Feb 15;142(4):233-9. doi: 10.7326/0003-4819-142-4-200502150-00005. PMID 15710956
- [Background] Doll R, Peto R, Boreham J, Sutherland I. Mortality in relation to smoking: 50 years' observations on male British doctors. BMJ. 2004 Jun 26;328(7455):1519. doi: 10.1136/bmj.38142.554479.AE. Epub 2004 Jun 22. PMID 15213107